CLINICAL TRIAL: NCT01970397
Title: A Prospective, Randomized, Controlled, Multi-center Study of the Safety and Effectiveness of JUVEDERM® Ultra XC Injectable Gel Versus Belotero Balance® for Perioral Lines
Brief Title: JUVEDERM® Ultra XC vs. Belotero Balance® for Perioral Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMA-JUV13001
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Results first posted 2015-09-02 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Patients With Moderate to Severe Perioral Lines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JUVEDERM® Ultra XC (Experimental): Perioral lines treated with JUVEDERM® Ultra XC
  Interventions: Device: JUVEDERM® Ultra XC
- Belotero Balance® (Experimental): Perioral Lines treated with Belotero Balance®
  Interventions: Device: Belotero Balance®

INTERVENTIONS:
Device: JUVEDERM® Ultra XC — Up to 3.0 mLs JUVEDERM® Ultra XC injected into the mid to deep dermis (2.0 mLs for initial treatment and 1.0 mL for touch-up treatment).
  Arms: JUVEDERM® Ultra XC
Device: Belotero Balance® — Up to 3.0 mLs Belotero Balance® injected into the mid to deep dermis (2.0 mLs for initial treatment and 1.0 mL for touch-up treatment).
  Arms: Belotero Balance®

SUMMARY:
A prospective, randomized, controlled, multi-center study of the safety and effectiveness of JUVEDERM® Ultra XC injectable gel versus Belotero Balance® for perioral lines

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe perioral lines as assessed by the Investigator using the 4-point POLSS (none, mild, moderate, and severe)
* Accept the obligation not to receive any other facial procedures or treatments at any time during the study that are not study related

Exclusion Criteria:

* Have lip tattoos, facial hair or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments
* Have dentures or any device covering all or part of the upper palate, and/or severe malocclusion, dentofacial or maxillofacial deformities, or significant asymmetry of the perioral area, as judged by the Treating Investigator
* Have a history of skin cancer
* Is an active smoker
* Has noticeable acne scarring, active inflammation, infection, cancerous or precancerous lesion, or unhealed wound in the mouth area
* Have had an active oral herpes or cold sore within 12 months
* Have undergone oral surgery or other dental procedures (e.g., tooth extraction, orthodontia, or implantation) within 30 days prior to enrollment or be planning to undergo any of these procedures during the study
* Have undergone cosmetic facial or perioral area procedures [e.g., face-lift, or other surgeries which may alter the appearance of the perioral area, including tissue grafting, or tissue augmentation with silicone, fat, or other permanent fillers] or be planning to undergo any of these procedures at any time during the study
* Have undergone temporary or semi-permanent facial dermal filler injections (e.g., hyaluronic acid, calcium hydroxylapatite, L-Polylactic acid) in the lower face (below the orbital rim) within 24 months
* Have received mesotherapy, or resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) within 6 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study other than study related procedures.
* Have begun use of any new over-the-counter or prescription, oral or topical, antiwrinkle products in the treatment area within 90 days prior to enrollment or be planning to begin use of such products at any time during the study. [NOTE: Use of sunscreens and continued therapy with some cosmeceuticals (e.g., alpha hydroxyl acids, glycolic acids, retinol, or retinoic acids) is allowed if the regimen was established ≥ 90 days prior to enrollment]
* Have had epilation (e.g. laser hair removal, electrolysis, threading, etc.) in the perioral area performed within 3 months
* Have received treatment with botulinum toxin of any serotype for any indication in the lower face [below the infraorbital rims (IORs)] within 1 year of the baseline visit

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2014-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Butterwick K, Marmur E, Narurkar V, Cox SE, Joseph JH, Sadick NS, Tedaldi R, Wheeler S, Kolodziejczyk JK, Gallagher CJ. HYC-24L Demonstrates Greater Effectiveness With Less Pain Than CPM-22.5 for Treatment of Perioral Lines in a Randomized Controlled Trial. Dermatol Surg. 2015 Dec;41(12):1351-60. doi: 10.1097/DSS.0000000000000576. PMID 26606435

RESULTS

PARTICIPANT FLOW:
Groups:
- JUVEDERM® Ultra XC: JUVEDERM® Ultra XC injected into perioral lines (2.0 mLs for initial treatment on Day 1 and 1.0 mL for touch-up treatment 2 weeks later if applicable).
- Belotero Balance®: Belotero Balance® injected into perioral lines (2.0 mLs for initial treatment on Day 1 and 1.0 mL for touch-up treatment 2 weeks later if applicable).
Period: Overall Study
Arm/Group | JUVEDERM® Ultra XC | Belotero Balance®
Started | 69 | 69
Completed | 67 | 64
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Personal Reasons | 1 | 2
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all randomized participants who received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | JUVEDERM® Ultra XC | Belotero Balance® | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (7.5) | 58.2 (9.26) | 58.2 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 68 | 135
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1 Point Improvement From Baseline on the Perioral Lines Severity Scale (POLSS)
Description: The investigator evaluated the severity of the participant's upper and low lip at Baseline (Pre-treatment) to Month 6 using the 4-point POLSS where None=No lines, Mild=Few, shallow lines, Moderate=Some, moderate lines or Severe=Many, deep lines or crevices. The percentage of participants with at least a 1 Point Improvement is reported.
Time Frame: Baseline, Month 6
Population: Participants from the Intent-to-treat population, all randomized treated participants, with data available for analysis at Month 6.
Measure: Number; unit: percentage of participants
Arm/Group | JUVEDERM® Ultra XC | Belotero Balance®
Number analyzed (Participants) | 67 | 65
percentage of participants | 87 | 72

2. Secondary Outcome: Participant Assessed Procedural and Post-Procedural Pain Levels
Description: The participant assessed procedural and post-procedural pain using an 11-point scale where: 0=no pain to 10=worst pain imaginable.
Time Frame: During injection, immediately following injection, 15, 30, and 45 min post-injection
Population: Intent-to-treat population included all randomized and treated participants.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | JUVEDERM® Ultra XC | Belotero Balance®
Number analyzed (Participants) | 68 | 68
units on a scale
  During Injection | 2.9 [2.4 to 3.5] | 4.4 [3.8 to 5.0]
  Immediately following Injection | 0.8 [0.5 to 1.1] | 1.8 [1.4 to 2.3]
  15 minutes following Injection | 0.1 [0.0 to 0.3] | 0.5 [0.3 to 0.7]
  30 minutes following Injection | 0.1 [0.0 to 0.2] | 0.3 [0.1 to 0.4]
  45 minutes following Injection | 0.0 [-0.0 to 0.1] | 0.2 [0.1 to 0.3]

3. Secondary Outcome: Subject's Global Assessment of Change in Appearance of Perioral Lines
Description: The participant evaluated the change in the appearance of their perioral lines (the lines that radiate outward from the edges of the upper and lower lips) using a 7-point scale where: 1 = Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse.
Time Frame: Baseline, Days 7, 14, Days 7, 14 after touch-up, Months 1, 3 and 6
Population: Participants from the Intent-to-treat population, all randomized treated participants, with data available at the given time-point.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | JUVEDERM® Ultra XC | Belotero Balance®
Number analyzed (Participants) | 68 | 68
units on a scale
  Day 7 | 1.8 [1.7 to 2.0] | 2.1 [1.9 to 2.2]
  Day 14 or Touch-up (n=66,67) | 1.7 [1.5 to 1.9] | 2.0 [1.8 to 2.2]
  Day 7 after Touch-up (n=30,42) | 1.6 [1.4 to 1.8] | 1.8 [1.6 to 2.0]
  Day 14 after Touch-up (n=32,40) | 1.8 [1.5 to 2.0] | 1.8 [1.6 to 2.0]
  Month 1 (n=66,67) | 1.7 [1.5 to 1.9] | 2.0 [1.8 to 2.1]
  Month 3 (n=68,65) | 1.8 [1.7 to 2.0] | 2.2 [2.0 to 2.4]
  Month 6 (n=67,65) | 1.9 [1.7 to 2.1] | 2.6 [2.3 to 2.8]

ADVERSE EVENTS:
Description: Safety population, all randomized treated participants, was used to determine the number of participants at risk for Serious and Non-serious adverse events.
Arm/Group | JUVEDERM® Ultra XC | Belotero Balance®
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 9/68 | 10/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JUVEDERM® Ultra XC (N=68) | Belotero Balance® (N=68)
Injection site bruise (General disorders) | 5 | 9
Injection site induration (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.